CLINICAL TRIAL: NCT04072458
Title: A Phase 1 Clinical Trial to Study the Safety, Pharmacokinetics, and Efficacy of BP1002 (L-Bcl-2) Antisense Oligonucleotide in Patients With Advanced Lymphoid Malignancies
Brief Title: A Clinical Trial of BP1002 in Patients With Advanced Lymphoid Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Path Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP1002-101-Lymph
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Mantle Cell Lymphoma; Peripheral T-cell Lymphoma (PTCL); Cutaneous T-cell Lymphoma (CTCL); Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); Follicular Lymphoma; Marginal Zone Lymphoma; Hodgkin Lymphoma; Waldenstrom Macroglobulinemia; DLBCL
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Hodgkin Disease; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BP1002 monotherapy (Experimental): L-Bcl-2 Antisense oligonucleotide (BP1002) is given in a sequential, dose escalation design. Starting dose is 20mg/m^2.
  Interventions: Drug: L-Bcl-2 antisense oligonucleotide

INTERVENTIONS:
Drug: L-Bcl-2 antisense oligonucleotide — There will be 2 planned dose levels, 20, and 40 mg/m^2. Successive cohorts of eligible patients with will be treated with BP1002. BP1002 is given as an intravenous infusion, twice weekly, as 8 doses per 28-day cycle. Cycles may be repeated every 4 weeks.
  Other Names: BP1002

SUMMARY:
This study evaluates the safety, pharmacokinetics, and efficacy of BP1002 (L-Bcl-2) antisense oligonucleotide in patients with advanced lymphoid malignancies. Up to 12 evaluable patients with a diagnosis of relapsed or refractory lymphoid malignancies are expected to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age
2. Patient has a life expectancy ≥ 3 month
3. Patient has relapsed or refractory disease Relapsed lymphoma: Relapsed lymphoma is disease that has responded to treatment but then returns.

   Refractory lymphoma: Failure to achieve complete response at the end of therapy or progression within 6 months from completion of therapy
4. Included Diseases

   * DLBCL, including transformed lymphoma
   * Mantle Cell Lymphoma
   * PTCL
   * CTCL
   * CLL/SLL
   * Follicular lymphoma
   * Marginal zone lymphoma
   * Hodgkin lymphoma (both classical and lymphocyte predominant)
   * Waldenströms Macroglobulinemia
5. Must has failed or is not a candidate for available therapies with reasonable likelihood of clinical benefit, which includes FDA approved products and standard of care regimens
6. Therapy means at least three front lines of therapy including Hematopoeitic Stem Cell Transplant (HSCT and/or Chimeric Antigen Receptor (CAR) T cells, when applicable
7. Females must be of non-childbearing potential, surgically sterile, postmenopausal, or practice adequate methods of contraception during the study
8. Males must agree to use an adequate method of contraception during the study
9. Eastern Cooperative Oncology Group (ECOG) Performance score of 0, 1, or 2
10. Adequate hepatic and renal functions as defined by:

    * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 times the upper limit of normal (ULN); and
    * Total bilirubin ≤1.5 times ULN; and
    * Estimated glomerular filtration rate (eGFR) of at least 50ml/min. These estimations can be calculated using the following methods:

      * Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation
      * Cockcroft Gault equation
      * Modification of Diet in Renal Disease (MDRD study equation)
      * Creatinine clearance estimated by 24-hr urine collection for creatinine clearance
11. Recovered from the effects of any prior surgery, radiotherapy, or antineoplastic treatment (with the exception of alopecia), based on Investigator assessment
12. Willing and able to provide written informed consent

Exclusion Criteria:

1. Active non-hematologic malignancy other than lymphoid malignancies treated with immuno- or chemotherapy within the previous 12 months except active non-melanoma, non-invasive skin cancer will be allowed
2. Known, active Central Nervous System (CNS) involvement of disease requiring intrathecal therapy. Note: Patients with a history of CNS disease may be allowed to participate based on at least 1 documented, negative spinal fluid assessment within 28 days prior to Screening
3. Patient eligible for high dose chemotherapy and autologous stem cell transplant
4. Indolent non-Hodgkin lymphoma (iNHL)
5. Patients at high risk of Tumor Lysis Syndrome (TLS)

   a. Bulky disease i. A unidimensional lesion greater than 10 cm and/or b. Lymphocyte count greater than 25,000 per µL
6. Receipt of any anti-cancer therapy within 14 days prior to Cycle 1 Day 1 (C1D1)
7. Uncontrolled active, untreated, or progressive infection
8. Receipt of any investigational agent or on study treatment within 30 days prior to C1D1
9. Females who are pregnant, test positive for pregnancy, or are breast-feeding during the Screening period, or intend to become pregnant or breast-feed during the course of the study or within 30 days after last dose of study drug
10. Serious intercurrent medical or psychiatric illness which, in the opinion of the Investigator, would interfere with the ability of the participant to complete the study
11. Active hepatitis B infection (based on positive surface antigen [HBsAg]), hepatitis C infection (based on Hepatitis C Virus (HCV) positive antibody [HCV Ab]), or human immunodeficiency virus (HIV-1 or HIV-2, based on positive antibody)
12. Presence of concurrent conditions that, in the opinion of the Investigator and/or Medical Monitor, may compromise or interfere with any aspect of study conduct or interpretation of results. This includes, but is not limited to, unstable or uncontrolled angina, New York Heart Association (NYHA) class III or IV congestive heart failure, uncontrolled and sustained hypertension, clinically significant cardiac dysrhythmia or clinically significant baseline EKG abnormality (e.g., QTcF >470 msec)
13. Within the past 6 months, has had any of the following: myocardial infarction, unstable angina pectoris, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack
14. Uncontrolled seizure disorder
15. Unable or unwilling to communicate or cooperate with the Investigator or follow the protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Identify Dose Limiting Toxicity (DLT) of BP1002 | 30 days
  Identify DLT of BP1002 using non-hematologic and hematologic measures per NCI CTCAE criteria
Identify and grade treatment-emergent adverse events (TEAE) of escalating doses of BP1002 | 30 days
  Identify TEAE of BP1002 using non-hematologic and hematologic measures per NCI CTCAE criteria
Identify and grade treatment-emergent laboratory abnormalities of escalating doses of BP1002 by identification and grading of | 30 days
  Identify and grade treatment-emergent laboratory abnormalities of BP1002 using non-hematologic and hematologic measures per NCI CTCAE criteria
Identify conduction and rhythm changes (treatment emergent QTc elevations or other treatment emergent changes in EKG intervals) of escalating doses of BP1002 | 30 days
  Collection of 12-lead EKGs at defined intervals to identify conduction and rhythm changes (treatment emergent QTc elevations or other treatment emergent changes in EKG intervals)
Recommended Phase 2 dose (RP2D) of BP1002 | 210 days
  Determine RP2D by evaluating Maximally Tolerated Dose (MTD) data: Any Dose Limiting Toxicity (DLT) observed will trigger an expansion of a cohort from 3 to 6 patients. A second DLT at any dose level will identify the Maximum Dose. The dose below that will be the MTD.
Determine plasma pharmacokinetics (PK) of BP1002 using maximum plasma drug concentration | 30 days
  Evaluate in vivo PK of BP1002 using maximum plasma drug concentration (Cmax)
Determine plasma pharmacokinetics (PK) of BP1002 using volume of distribution | 30 days
  Evaluate in vivo PK of BP1002 volume of distribution (Vd)
Determine plasma pharmacokinetics (PK) of BP1002 using elimination rate constant | 30 days
  Evaluate in vivo PK of BP1002 elimination rate constant
Determine half-life plasma pharmacokinetics (PK) of BP1002 | 30 days
  Evaluate in vivo PK of BP1002 half-life (t1/2)
Determine pharmacokinetics (PK) of BP1002 | 30 days
  12-lead EKG assessments will be collected and analyzed for conduction and rhythm changes (treatment emergent QTc elevations or other treatment emergent changes in EKG intervals) from those the EKG obtained immediately before the first BP1002 dose, and after BP1002 dose, and will mirror the time points used to collect the plasma PK assessments

SECONDARY OUTCOMES:
Determine evidence of tumor response by bone marrow aspirate | 30 days
  Assess tumor response by evaluating bone marrow aspirate to determine complete response (CR), partial response (PR), or minor response (MR) using appropriate uniform response criteria as published by Response Evaluation Criteria in Lymphoma (RECIL) 2017, CLL guidelines, and International Workshop on Waldenström's Macroglobulinemia (IWWM 6th)
Determine evidence of tumor response by Complete Blood Count (CBC) | 30 days
  Assess tumor response by evaluating CBC measurements to determine complete response (CR), partial response (PR), or minor response (MR) using appropriate uniform response criteria as published by Response Evaluation Criteria in Lymphoma (RECIL) 2017, CLL guidelines, and International Workshop on Waldenström's Macroglobulinemia (IWWM 6th)
Determine estimates for time to progression (TTP) | 30 days
  Measured from treatment start date to date of progression by CBC and/or bone marrow aspirate
Determine estimates for progression-free survival (PFS) | 30 days
  Measured from treatment start date to date of progression or death by CBC and/or bone marrow aspirate
Determine estimates for event-free survival (EFS) | 30 days
  Measured from treatment start date to date of progression, death, or change in therapy by CBC and/or bone marrow aspirate
Activity of BP1002 on Bcl-2 expression in tumor samples | 30 days
  Flow cytometric assays to determine the effects of BP1002 on Bcl-2 protein expression using patient blood samples

OTHER OUTCOMES:
Exploratory objective to correlate treatment response with cytogenetic characteristics | 30 days
  Flow cytometric assays to determine the effects of BP1002 on Bcl-2 protein expression
Exploratory objective to correlate treatment response with molecular characteristics | 30 days
  Flow cytometric assays to determine the effects of BP1002 on Bcl-2 protein expression

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Georgia Cancer Center, Augusta, Georgia
  - New York Medical College / Westchester Medical Center, Valhalla, New York
  - Sarah Cannon Research Institute/Tennesee Oncology, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Research Center, Houston, Texas